CLINICAL TRIAL: NCT03503409
Title: A Single-arm Phase II Multicenter Study of IDH1 (AG 120) Inhibitor in Patients With IDH1 Mutated Myelodysplastic Syndrome
Brief Title: IDH1 (AG 120) Inhibitor in Patients With IDH1 Mutated Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIOME-STUDY
Record Dates: First submitted 2018-04-04; First posted 2018-04-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — ivosidenib

STUDY DESIGN:
Intervention Model Description: Subjects enrolled will receive continuous 28-day cycles of AG-120. AG-120 will be dispensed on Day 1 of each treatment cycle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AG-120 (Experimental): Subjects enrolled will receive continuous 28-day cycles of AG-120 - 500 mg. AG-120 will be dispensed on Day 1 of each treatment cycle
  Interventions: Drug: AG-120

INTERVENTIONS:
Drug: AG-120 — 500 mg/day Oral of AG-120. AG-120 will be dispensed on Day 1 of each treatment cycle

SUMMARY:
patients with MDS (Myelodysplastic Syndrome) and mutated IDH1 patients will be treated with AG120 (IDH1 inhibitor)

DETAILED DESCRIPTION:
Myelodysplastic syndrome (MDS) are clonal hematopoietic stem cell disorders characterized by ineffective hematopoiesis leading to blood cytopenia, especially anemia, and often evolving to Acute myeloblastic Leukemia (AML). Main prognostic factors of MDS, for progression to AML and survival, include the number and importance of cytopenias, percent marrow blasts and bone marrow cytogenetic abnormalities. These factors are combined in an International Prognostic Scoring System (IPSS) that distinguishes 4 subgroups with significantly different risk of progression to AML and survival (low, intermediate 1 (int 1), intermediate 2 (int 2), high). Low and int 1 subgroups are often grouped together as "favorable " or low risk MDS, and int 2 and high subgroups are " unfavorable " or high risk MDS.

On the other hand, only 50 to 60% of the patients respond to Azacitidine, and most responders relapse within 12 to 15 months resulting in a median survival of only about 6 months in these patients,. As a result there is a need for new therapies in patients who fail to respond to azacitidine or decitabine and for whom there is currently no establish treatment.

Isocitrate dehydrogenase 1 and 2 (IDH1 and IDH2) are key metabolic enzymes that convert isocitrate to α-ketoglutarate. IDH1/2 mutations define distinct subsets of cancers, including low-grade gliomas and secondary glioblastomas, chondrosarcomas, intrahepatic chol- angiocarcinomas, and hematologic malignancies. Somatic point mutations in IDH1/2 confer a gain-of-function in cancer cells, resulting in the accumulation and secretion in vast excess of an oncometabolite, the D-2-hydroxyglutarate (D-2HG). Overproduction of D-2HG interferes with cellular metabolism and epigenetic regulation, contributing to oncogenesis. Indeed, high levels of D-2HG inhibit alpha-ketoglutarate-dependent dioxygenases, including histone and DNA demethylases, leading to histone and DNA hypermethylation and finally a block in cell differentiation.

preclinical studies have demonstrated that inhibition of IDH1/2-mutant enzymes decreases intracellular D-2-hydroxyglutarate (D-2HG) levels, reverses epigenetic dysregulation, and releases the differentiation block.

AG-120, a selective inhibitor of the IDH1 mutant enzyme Overall, in myeloid malignancies, AG120 have been mainly used in generally heavily pretreated AML, with about 40% of responses in patients with the respective IDH 1 mutation, and a median response duration exceeding 1 year when CR or PR was achieved.

Based on these results, we hypothesize that the IDH1 inhibitor (AG 120) may be an effective therapeutic option in patient with IDH1 mutation-positive myelodysplastic syndrome This is an open-label, single-arm multicenter, phase II study

The efficacy of AG 120 will be studied in 3 different groups of MDS patients with IDH-1 mutation:

* Cohort A: Higher risk MDS without response (Complete response (CR), Partial Response (PR) ,stable disease with HI) after at least 6 cycles of azacitidine or relapse after a response
* Cohort B: Untreated higher risk MDS without life threatening cytopenias (ie Absolute neutrophil count (ANC )< 500/mm3 or any recent infection, platelets below 30,000/mm3 or any bleeding symptom). Azacitidine will be added after 3 cycles of AG 120 in the absence of significant IWG 2006 criteria response
* Cohort C: Lower risk MDS with anemia resistant to erythropoietic stimulating agents (primary or secondary resistance)

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to participate in the study:
* Age ≥ 18 years
* Myelodysplastic syndrome according to WHO classification including non-proliferative AML up to 29% of BM blast
* Belonging to one of the following categories :
* higher risk (IPSS high or int 2 ) MDS without response to azacitidine (CR,PR, stable disease with HI) after at least 6 cycles , or relapsing after a response but without overt progression (defined by at least doubling of marrow blasts, compared to pre azacitidine bone marrow, or AML progression beyond 30% blasts)
* Untreated higher risk MDS (IPSS int-2, high) without life threatening cytopenia including ANC <500/mm3 or any recent severe infections and /or platelets below 30,000/mm3 or any bleeding symptom
* lower risk MDS with resistance or loss of response to a previous treatment with epoetin alpha/ beta (≥60000 U/w) or Darbopoetin (≥250 ug/w) given for at least 12 weeks and RBC transfusion requirement at least 2 U/8 weeks in the previous 16 weeks
* Presence of IDH1 mutation in either blood or marrow prior to start of therapy;
* Normal renal function, defined by creatinine less than 1.5 times the upper limit of normal, creatinine clearance (Modification of diet in renal disease) creatinine clearance ≥ 50 mL/min;
* Normal liver function, defined by total bilirubin and transaminases less than 1.5 times the upper limit of normal;
* Adequate cardiac ejection fraction (>40%);
* Patient is not known to be refractory to platelet transfusions;
* Written informed consent;
* Patient must understand and voluntarily sign consent form.
* Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements;
* ECOG performance status 0-2 at the time of screening;
* Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy. Subjects with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 3 months (females and males) following the last dose of AG-120. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices.
* Male patients must :

  * Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment.
  * Agree to learn about the procedures for preservation of sperm before starting treatment

Exclusion Criteria:

* A patient meeting any of the following criteria is not eligible to participate in the study:
* Severe infection or any other uncontrolled severe condition.
* Significant cardiac disease - NYHA Class III or IV or having suffered a myocardial infarction in the last 6 months.
* Less than 14 days since prior treatment with growth factors (EPO, G-CSF).
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before the study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicity from any previous therapy.
* Subject has a heart-rate corrected QT interval using Fridericia's method (QTcF) ≥ 470 msec or any other factor that increases the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with prolonged QTcF interval in the setting of bundle branch block may participate in the study.
* Subject is taking known strong cytochrome P450 (CYP) 3A4 inducers or inhibitors or sensitive CYP3A4 substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
* Subject is taking P-glycoprotein (P-gp) transporter-sensitive substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within ≥ 5 half-lives prior to administration of study treatment
* Active cancer or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast.
* Patient already enrolled in another therapeutic trial of an investigational drug.
* Known HIV infection or active hepatitis B or C.
* Women who are or could become pregnant or who are currently breastfeeding.
* Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form.
* Patient eligible for allogeneic stem cell transplantation.
* Known allergies to AG 120 or any of its excipients.
* The study does not provide for the inclusion of persons referred to in Articles L. 1121-5 to L. 1121-9 and L. 1122-1-2 of the Public Health Code (e.g. minors, protected adults, etc.)
* No affiliation to a health insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2027-04-02 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
Overall hematological response | 6 months
  overall hematological response

SECONDARY OUTCOMES:
response duration | 3 years
  response duration
IPSS progression | 3 years
  time to IPSS progression

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sébert, Dr, Principal Investigator — APHP
Locations (38):
- France (25):
  - CH Angers, Angers
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hôpital Nord Franche-Comté/Service de médecine interne / Hématologie clinique, Belfort
  - CHU côte de Nacre, Caen
  - CHU de Grenoble/Clinique Universitaire d'hématologie 6e A, Grenoble
  - CH Le Mans/Service d'hématologie Oncologie, Le Mans
  - CHRU de Limoges, Limoges
  - centre hospitalier de Lyon, Lyon
  - Institut Paoli Calmettes/Unité d'Hématologie 3, Marseille
  - CHU Montpellier St Eloi, Montpellier
  - Hôpital E. Muller-GHR Mulhouse Sud-Alsace, Mulhouse
  - CHU Hôtel Dieu/Service d'Hématologie Clinique, Nantes
  - Hôpital Archet 1/Service d'Hématologie Clinique, Nice
  - GHU Caremeau, Nîmes
  - Hôpital Saint Louis - Hématologie Séniors, Paris
  - Hôpital Necker, Paris
  - Hôpital Henri Mondor, Paris
  - CHU de Haut-Lévèque/Centre François Magendie/Service des maladies du sang, Pessac
  - CHU de Poitiers/Pôle de cancérologie - secteur tertiaire-, Poitiers
  - Centre Henri Becquerel, Rouen
  - institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Médecine Interne/IUCT Oncopole, Toulouse
  - CHU de Tours, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier de Versailles-Hôpital André Mignot, Versailles
- Italy (13):
  - Ematologia ALESSANDRIA, Alessandria
  - CLINICA Ematologica ANCONA, Ancona
  - Ematologia BOLOGNA, Bologna
  - Ematologia BRESCIA, Brescia
  - Ematologia FIRENZE, Florence
  - Clinica Ematologica Genova, Genova
  - Ematologia GENOVA, Genova
  - Ematologia LECCE, Lecce
  - Ematologia MILANO, Milan
  - Ematologia ORBASSANO, Orbassano
  - Ematologia ed Immunologia Clinica PADOVA, Padua
  - Reggio Calabria, Reggio Calabria
  - Ematologia ROMA, Roma

IPD SHARING:
Plan to Share IPD: No